CLINICAL TRIAL: NCT05315206
Title: Modulation of Neuronal Connettivity Along the Visual Pathways in Patients Affected by Glaucoma Throug Treatment With Citicoline Oral Solution: Multimodal Morpho-funcional Study
Brief Title: Multimodal Morpho-functional Study in Glaucoma Patients-Citicoline Oral Solution
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione G.B. Bietti, IRCCS (Other)
Responsible Party: Principal Investigator, Dr. Vincenzo Parisi, Head of Neurophysiology and Neurophthalmology Research Unit, Fondazione G.B. Bietti, IRCCS
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 128/21/FB
Record Dates: First submitted 2022-02-04; First posted 2022-04-07 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Primary Open Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Cytidine Diphosphate Choline

STUDY DESIGN:
Intervention Model Description: Patients selected according to the inclusion / exclusion criteria, after signing the informed consent, will be randomized into two groups:
  1. In a group of patients with open angle glaucoma (OAG), Citicoline in oral solution (10 ml / day, Neurotidine®) will be administered for 12 months (Citicoline Treated Group, TC Group)
  2. in another group of patients with OAG will be administered Placebo (Containing all excipients of Neurotidine ®) (10 ml / day) for 12 months (Placebo Treated Group, TP Group)
Who Masked: Participant, Care Provider, Investigator
Masking Description: Only after the signing of the informed consent, a single investigator ("enrolling physician"), not involved in the clinical and instrumental evaluations, will decide whether to assign the selected patient to one of two groups: treated-Citicoline or treated-Placebo.
  Randomization will be done by dividing the selected patients into two groups based on similar characteristics of: age, perimetric defect and, mainly,retinal cortical time (RCT) values.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Citicoline Treated Group, TC Group (Experimental): In a group of patients with open angle glaucoma (OAG), Citicoline in oral solution (10 ml / day) will be administered for 12 months (Citicoline Treated Group, TC Group)
  Interventions: Dietary Supplement: Citicoline
- Placebo Treated Group, TP Group (Placebo Comparator): in another group of patients with open angle glaucoma (OAG) will be administered Placebo (Containing all excipients of Citicoline in oral solution) (10 ml / day) for 12 months (Placebo Treated Group, TP Group)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Citicoline — The patient will be given 10 ml of Citicoline oral solution (Neurotidine ®) once a day in the morning for 1 year. To patients will be given 4 bottles containing 500 ml of Citicoline and the relative instructions for administration. After 6 months, the patient will bring back the used bottles and will be given additional 4 bottles containing Citicoline (Neurotidine ®). Again at the end of this 6 month period the patient will bring back the used bottles.
  Each bottle of Neurotidine will contain: water; fructose; Citicoline (500 mg per 10 ml); acidity regulators: sodium citrate, sodium hydroxide; preservative: potassium sorbate; dye: riboflavine.
  Arms: Citicoline Treated Group, TC Group
Dietary Supplement: Placebo — The patient will be given 10 ml of an oral solution of Placebo. Each bottle of Placebo, the solution of which will be indistinguishable from the active product in terms of appearance and flavor, will contain: water; fructose; acidity regulators: sodium citrate, sodium hydroxide; preservative: potassium sorbate; dye: riboflavin
  Arms: Placebo Treated Group, TP Group

SUMMARY:
A prospective, multicentre, randomized, blinded, masked study that involves the enrollment of 60 patients affected by open angle glaucoma (OAG).

Patients selected according to the inclusion / exclusion criteria, after signing the informed consent, will be randomized into two groups:

1. In a group of patients with OAG, Citicoline in oral solution (10 ml / day, Neurotidine®) will be administered for 12 months (Citicoline Treated Group, TC Group)
2. in another group of patients with OAG will be administered Placebo (Containing all excipients of Neurotidine ®) (10 ml / day) for 12 months (Placebo Treated Group, TP Group) Randomization will be done by dividing the selected patients into two groups based on similar characteristics of: age, perimetric defect and, mainly, retinal-cortical time (RCT) values.

Patients will be assigned to each group by an investigator not involved in functional and structural testing.

The key will be opened only at the end of the treatment in order to evaluate the first effects.

The Primary Objective was to evaluate whether treatment with Citicoline in oral solution can produce an improvement of the post-retinal neural conduction, that is delayed in patients with OAG.

The Secondary objective was to evaluate in patients with OAG whether the possible changes in post-retinal neural conduction induced by treatment with Citicoline in oral solution (information obtained through electrophysiological recordings) are associated or not with morphological and functional variations of the nervous structures forming the visual pathways (nucleus geniculatus lateral, optic tract, visual cortex, information obtained through the acquisition of structural and functional magnetic resonance imaging) and whether both conditions can be related to the morpho-functional variations of the retinal ganglion cells and of the visual field (VF).

DETAILED DESCRIPTION:
Sixty patients affected by bilateral open angle glaucoma, between the ages of 20 and 70, will be enrolled in the study within a maximum time frame of 12 months. The enrollment will be performed at T0 (screening), in this occasion an extensive ophthalmological evaluation will be performed after the signature of the informed consent. The patient will be undergoing to the evaluation of Best corrected Visual Acuity (BCVA), intraocular pressure (IOP), fundus examination, Visual Field (VF) exam (Humphrey 24-2and 10-2 standard SITA) Visual Evoked Potentials (VEP) and pattern electroretinogram (PERG). Moreover a morphological examination of optic nerve and macular area was assessed by Optical Coherence Tomography (OCT) with the analysis of retinal nerve fiber layer (RNFL) and retinal ganglion cells (RGCs).

Patients included in the study present a Mean Deviation defect (MD), tested at the VF examination, between -6 and -25 dB and an increase in Retinal-Cortical Time (RCT) response. RCT is a measure derived through the difference of Implicit Time values of latency of simultaneous recording of visual evoked potential (VEP) and pattern electroretinogram (PERG), which represent a post-retinal nerve conduction delay.

About 7-15 days after T0 a new ophthalmological examination will be performed (T1). The patient will be undergoing to the evaluation of BCVA, IOP, fundus examination, VF exam (Humphrey 24-2and 10-2 standard SITA), VEP, PERG and OCT. In this occasion a Magnetic Resonance Imaging (MRI) of the brain will be performed.

At the end of this evaluation, the patient will be given 4 bottles containing 500 ml of Citicoline in oral solution (Neurotidine®) or Placebo and will be given the relative instructions for administration. The posology will be 10 ml once a day in the morning for 6 months. At the end of the 6 month period the patient will be asked to hand over the used bottles.

After 6 months ± 10 days, a novel complete ophthalmologic evaluation will be performed (T2) (BCVA, IOP, VF exam, VEP, PERG, OCT), and patients will be given an additional 4 bottles containing Neurotidine ® or Placebo and will be given instructions for their administration. Again at the end of this 6 month period the patient will bring back the used bottles.

One year after T0, a last complete ophthalmological visit (BCVA, IOP, VF exam, VEP, PERG, OCT) will be performed (T3). In this visit MRI will be repeated. At the end of the visit, the patient will bring back the used bottles. Will be asked to the patient if adverse events will occurs during such period.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 70 years old
* Diagnosis of glaucoma. Glaucoma is defined as: glaucomatous damage of the CV (Humphrey 24-2 standard SITA with mean deviation between -6 and -25 dB) and glaucomatous appearance of the optic nerve
* Visual acuity not less than 5/10
* Eye pressure below 21 mmHg with the use of ocular hypotonizing drugs including sympathomimetics, beta-blockers, prostaglandins, beta-adrenergics, carbonic anhydrase inhibitors. Such drugs can be used both alone and in combination with each other.
* Documented post-retinal nerve conduction delay through simultaneous recording of VEP and PERG showing an increase in RCT

Exclusion Criteria:

* Ocular surgery in the 3 months preceding the study, including surgery for cataracts in the previous three months.
* Cataract or maculopathy
* Argon laser trabeculoplasty (ALT) within the previous 6 months
* Known hypersensitivity to the study product
* Secondary causes of ocular hypertension, including systemic or topical use of steroids
* Positive history of ocular or systemic diseases that could preclude enrollment in the study in the opinion of the investigators
* Changes in systemic therapies that could compromise intraocular pressure values (beta-blockers, alpha and beta adrenergics, calcium inhibitors, ACE inhibitors) in the 30 days prior to enrollment
* Ongoing therapy with vasoactive cerebral drugs, neurotrophic, lutein, zeaxanthin, retinal, acid, docosahexaenoic, Ubiquinone and / or its derivatives, Citicoline and / or its derivatives (possible previous treatment with Ubiquinone, L-Carnitine, Citicoline and / or its derivatives must have been suspended at least 6 months prior to inclusion in the study)
* Pregnancy, breastfeeding
* Diabetes
* Systemic lupus erythematosus, rheumatoid arthritis, connectivitis
* Concomitant use of anticoagulants and lithium

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2022-01-25 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Retino-cortical time (RCT) changes after treatment with citicoline in oral solution. | One year
  The changes of the retino-cortical time (RCT) in patients affected by open angle glaucoma after one years of treatment with Citicoline in oral solution compared to patients affected by open angle glaucoma treated with placebo.

SECONDARY OUTCOMES:
Correlation between RCT changes and morpho-functional parameters changes after treatment with citicoline in oral solution. | one year
  In patients with open angle glaucoma, the changes of retino-cortical time (RCT) are associated or not with morphological and functional changes in the nerve structures that form the optical pathways, measured by OCT (RNFL and RGCs), visual field (MD) and magnetic resonance, after one year of treatment with Citicoline in oral solution respect to patients treated with Placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo VP Parisi, MD, Principal Investigator — IRCSS Fondazione Bietti
Locations (2):
- Italy (2):
  - Fondazione BIetti, Britannico Hospital, Roma
  - Fondazione G.B. Bietti-IRCCS, Rome

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: As soon as possible when the study will be completed. About 6 months after the end of the data collection
Access Criteria: The results of this study will be avaiable after end of the study ( 18-24 months) and their publication on a scientific journal.

REFERENCES:
- [Result] Quigley HA, McKinnon SJ, Zack DJ, Pease ME, Kerrigan-Baumrind LA, Kerrigan DF, Mitchell RS. Retrograde axonal transport of BDNF in retinal ganglion cells is blocked by acute IOP elevation in rats. Invest Ophthalmol Vis Sci. 2000 Oct;41(11):3460-6. PMID 11006239
- [Result] Lipton SA, Rosenberg PA. Excitatory amino acids as a final common pathway for neurologic disorders. N Engl J Med. 1994 Mar 3;330(9):613-22. doi: 10.1056/NEJM199403033300907. No abstract available. PMID 7905600
- [Result] Oddone F, Lucenteforte E, Michelessi M, Rizzo S, Donati S, Parravano M, Virgili G. Macular versus Retinal Nerve Fiber Layer Parameters for Diagnosing Manifest Glaucoma: A Systematic Review of Diagnostic Accuracy Studies. Ophthalmology. 2016 May;123(5):939-49. doi: 10.1016/j.ophtha.2015.12.041. Epub 2016 Feb 15. PMID 26891880
- [Result] Parisi V. Impaired visual function in glaucoma. Clin Neurophysiol. 2001 Feb;112(2):351-8. doi: 10.1016/s1388-2457(00)00525-3. PMID 11165541
- [Result] Burgoyne CF, Downs JC, Bellezza AJ, Suh JK, Hart RT. The optic nerve head as a biomechanical structure: a new paradigm for understanding the role of IOP-related stress and strain in the pathophysiology of glaucomatous optic nerve head damage. Prog Retin Eye Res. 2005 Jan;24(1):39-73. doi: 10.1016/j.preteyeres.2004.06.001. PMID 15555526
- [Result] Furlanetto RL, Teixeira SH, Gracitelli CPB, Lottenberg CL, Emori F, Michelan M, Amaro E Jr, Paranhos A Jr. Structural and functional analyses of the optic nerve and lateral geniculate nucleus in glaucoma. PLoS One. 2018 Mar 23;13(3):e0194038. doi: 10.1371/journal.pone.0194038. eCollection 2018. PMID 29570721
- [Result] Schmidt MA, Knott M, Heidemann R, Michelson G, Kober T, Dorfler A, Engelhorn T. Investigation of lateral geniculate nucleus volume and diffusion tensor imaging in patients with normal tension glaucoma using 7 tesla magnetic resonance imaging. PLoS One. 2018 Jun 7;13(6):e0198830. doi: 10.1371/journal.pone.0198830. eCollection 2018. PMID 29879191
- [Result] Aksoy DO, Umurhan Akkan JC, Alkan A, Aralasmak A, Otcu Temur H, Yurtsever I. Magnetic Resonance Spectroscopy Features of the Visual Pathways in Patients with Glaucoma. Clin Neuroradiol. 2019 Dec;29(4):615-621. doi: 10.1007/s00062-018-0728-7. Epub 2018 Oct 5. PMID 30291364
- [Result] Wang Y, Wang X, Zhou J, Qiu J, Yan T, Xie Y, Li L, Lu W. Brain morphological alterations of cerebral cortex and subcortical nuclei in high-tension glaucoma brain and its associations with intraocular pressure. Neuroradiology. 2020 Apr;62(4):495-502. doi: 10.1007/s00234-019-02347-1. Epub 2019 Dec 23. PMID 31872278
- [Result] Gracitelli CPB, Duque-Chica GL, Sanches LG, Moura AL, Nagy BV, Teixeira SH, Amaro E Jr, Ventura DF, Paranhos A Jr. Structural Analysis of Glaucoma Brain and its Association With Ocular Parameters. J Glaucoma. 2020 May;29(5):393-400. doi: 10.1097/IJG.0000000000001470. PMID 32079996
- [Result] Parisi V, Manni G, Colacino G, Bucci MG. Cytidine-5'-diphosphocholine (citicoline) improves retinal and cortical responses in patients with glaucoma. Ophthalmology. 1999 Jun;106(6):1126-34. doi: 10.1016/S0161-6420(99)90269-5. PMID 10366081
- [Result] Parisi V, Centofanti M, Ziccardi L, Tanga L, Michelessi M, Roberti G, Manni G. Treatment with citicoline eye drops enhances retinal function and neural conduction along the visual pathways in open angle glaucoma. Graefes Arch Clin Exp Ophthalmol. 2015 Aug;253(8):1327-40. doi: 10.1007/s00417-015-3044-9. Epub 2015 May 26. PMID 26004075
- [Result] Parisi V. Electrophysiological assessment of glaucomatous visual dysfunction during treatment with cytidine-5'-diphosphocholine (citicoline): a study of 8 years of follow-up. Doc Ophthalmol. 2005 Jan;110(1):91-102. doi: 10.1007/s10633-005-7348-7. PMID 16249960
- [Result] Parisi V, Coppola G, Centofanti M, Oddone F, Angrisani AM, Ziccardi L, Ricci B, Quaranta L, Manni G. Evidence of the neuroprotective role of citicoline in glaucoma patients. Prog Brain Res. 2008;173:541-54. doi: 10.1016/S0079-6123(08)01137-0. PMID 18929133
- [Result] Parisi V, Barbano L, Di Renzo A, Coppola G, Ziccardi L. Neuroenhancement and neuroprotection by oral solution citicoline in non-arteritic ischemic optic neuropathy as a model of neurodegeneration: A randomized pilot study. PLoS One. 2019 Jul 26;14(7):e0220435. doi: 10.1371/journal.pone.0220435. eCollection 2019. PMID 31348806
- [Result] Parisi V, Oddone F, Ziccardi L, Roberti G, Coppola G, Manni G. Citicoline and Retinal Ganglion Cells: Effects on Morphology and Function. Curr Neuropharmacol. 2018;16(7):919-932. doi: 10.2174/1570159X15666170703111729. PMID 28676014
- [Result] Oddone F, Rossetti L, Parravano M, Sbardella D, Coletta M, Ziccardi L, Roberti G, Carnevale C, Romano D, Manni G, Parisi V. Citicoline in Ophthalmological Neurodegenerative Disease: A Comprehensive Review. Pharmaceuticals (Basel). 2021 Mar 20;14(3):281. doi: 10.3390/ph14030281. PMID 33804675
- [Result] Rejdak R, Toczolowski J, Kurkowski J, Kaminski ML, Rejdak K, Stelmasiak Z, Grieb P. Oral citicoline treatment improves visual pathway function in glaucoma. Med Sci Monit. 2003 Mar;9(3):PI24-8. PMID 12640353
- [Result] Virno M, Pecori-Giraldi J, Liguori A, De Gregorio F. The protective effect of citicoline on the progression of the perimetric defects in glaucomatous patients (perimetric study with a 10-year follow-up). Acta Ophthalmol Scand Suppl. 2000;(232):56-7. doi: 10.1111/j.1600-0420.2000.tb01107.x. No abstract available. PMID 11235540
- [Result] Roberti G, Tanga L, Parisi V, Sampalmieri M, Centofanti M, Manni G. A preliminary study of the neuroprotective role of citicoline eye drops in glaucomatous optic neuropathy. Indian J Ophthalmol. 2014 May;62(5):549-53. doi: 10.4103/0301-4738.133484. PMID 24881599
- [Result] Parisi V, Gallinaro G, Ziccardi L, Coppola G. Electrophysiological assessment of visual function in patients with non-arteritic ischaemic optic neuropathy. Eur J Neurol. 2008 Aug;15(8):839-45. doi: 10.1111/j.1468-1331.2008.02200.x. Epub 2008 Jun 28. PMID 18557920
- [Result] Parisi V, Miglior S, Manni G, Centofanti M, Bucci MG. Clinical ability of pattern electroretinograms and visual evoked potentials in detecting visual dysfunction in ocular hypertension and glaucoma. Ophthalmology. 2006 Feb;113(2):216-28. doi: 10.1016/j.ophtha.2005.10.044. Epub 2006 Jan 10. PMID 16406535

DOCUMENTS (2):
  • Study Protocol (2021-10-15): https://cdn.clinicaltrials.gov/large-docs/06/NCT05315206/Prot_000.pdf
  • Informed Consent Form (2021-10-15): https://cdn.clinicaltrials.gov/large-docs/06/NCT05315206/ICF_001.pdf